CLINICAL TRIAL: NCT04195724
Title: Microbiome Translocation in Different Circulatory Compartments in Decompensated Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Jinjun Chen, Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Cirrhosis, Liver
Keywords: gut microbial translocation; metagenomic next-generation sequencing; transjugular intrahepatic portosystemic shunt
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with decompensated ascites and receiving TIPS (Experimental): Patients with decompensated ascites and receiving TIPS will be enrolled. In this study, diagnostic paracentesis will be performed to get the ascites sample before the patients receiving TIPS. Next, the blood sample from superior mesenteric vein and hepatic vein will be collected under the procedure of TIPS.
  Interventions: Other: mNGS for pathogen detection

INTERVENTIONS:
Other: mNGS for pathogen detection — mNGS for pathogen detection and metabonomics (ascites, fecal,venous blood from superior mesenteric vein, hepatic vein and peripheral vein, respectively)

SUMMARY:
Acquired dysfunctional immunity in cirrhosis predisposes patients to frequent bacterial infections contributing to disease progression and may lead to the development of acute-on-chronic liver failure (ACLF). Spontaneous bacterial peritonitis (SBP) is one of the most frequent infections in cirrhosis and therefore a trigger for ACLF. ACLF is characterized by systemic inflammation even in the absence of confirmed infection and associated with poor outcome. The source of ascites infection, especially in case of culture-positive SBP and bacterascites, is suspected to be bacterial translocation from gut.

In decompensated cirrhosis, data on the gut microbial translocation in different circulatory compartments is limited. Moreover, the link between gut microbiome and systemic inflammation in liver disease has still not established.

The transjugular intrahepatic portosystemic shunt (TIPS) is applied to treat portal hypertension which frequently leads to intestinal bleeding, life-threatening esophageal bleeding and ascites. Under the procedure of TIPS, the vein blood samples in different compartments (superior mesenteric vein, portal vein and hepatic vein) from patients with decompensated liver cirrhosis are available. Metagenomic next-generation sequencing (mNGS) is a promise approach for the diagnosis of infectious disease because a comprehensive spectrum of potential causes (viral, bacterial, fungal, and parasitic) can be identified by a single assay. Previous study reported that mNGS of cerebrospinal fluid can be applied to diagnosis of meningitis and encephalitis. Comparing to traditional bacterial culture method, mNGS method is more sensitive and rapidly in pathogen detection. Therefore, the circulating microbiome in different compartment can be characterized by means of mNGS.

Here, the study aim to investigate the circulating microbiome from superior mesenteric vein (first venous outflow in gut-liver axis), hepatic vein (liver outflow), peripheral vein and ascites from patients with decompensated liver cirrhosis receiving TIPS. Before TIPS, fecal sample and unary sample are collected. And mNGS method is performed to identify the pathogen in ascites,fecal and blood samples in a single center. Ultimately, the study aim to build up the link between gut microbiome translocation and liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years old;
2. Patients with decompensated liver cirrhosis;
3. Patients receiving TIPS for either variceal bleeding or refractory ascites.

Exclusion Criteria:

1. Hepatic tumor or extrahepatic related cancer;
2. Not provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The circulating microbiome in ascites,fecal and in blood of different circulatory compartments (superior mesenteric vein, peripheral vein and hepatic vein, respectively). | 28 days
  mNGS and metabonomics are performed in ascites,fecal and in blood of different circulatory compartments (superior mesenteric vein, peripheral vein and hepatic vein, respectively).

SECONDARY OUTCOMES:
The improvement of gut microbiome translocation 6 months after the operation of TIPS. | 6 months after discharge
  The improvement of gut microbiome translocation 6 months is evaluated after the operation of TIPS.
The occurrence of decompensated events (infection, ascites, hepatic encephalopathy, gastrointestinal bleeding) 1 year after the operation of TIPS. | 1 years after discharge
  The occurrence of decompensated events are recorded during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jinjun Chen, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China